CLINICAL TRIAL: NCT06150794
Title: Intra-matrical Methotrexate Alone Versus Its Combination With Excimer Light in Treatment of Nail Psoriasis
Brief Title: Methotrexate Alone vs Combination With Excimer Light in Nail Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manar Elammary, Investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASU-MTX
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Nail Psoriasis
Keywords: Nail psoriasis; chronic psoriasis; methotrexate; excimer laser
MeSH Terms: interventions — Lasers, Excimer; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTX alone (arm 1) (Active Comparator): Participants will receive intra-matrical methotrexate injection in the affected fingers of both hands, once a month for 3 months.
  Comparison arms represent right hand (MTX+EL) and left hand (MTX alone) in the same participants.
  Interventions: Drug: Methotrexate Injection
- MTX + EL (arm 2) (Active Comparator): Participants will receive excimer laser treatment in the affected fingers of the right hand only, in addition to treatment with methotrexate injection the same participants are receiving in the same hand.
  Excimer laser will be applied twice weekly for 3 months.
  Comparison arms represent right hand (MTX+EL) and left hand (MTX alone) in the same participants.
  Interventions: Device: Excimer laser; Drug: Methotrexate Injection

INTERVENTIONS:
Device: Excimer laser — Excimer laser will be started at a dose of 300 mj/cm2 and increases 50-100 mj/cm2 each session. The aim of treatment is to deliver a dose that induces visible redness in the psoriatic lesion (supra-erythematous dose), but not induce a blister.
  Arms: MTX + EL (arm 2)
Drug: Methotrexate Injection — A ring block with 0.5 mL plain lignocaine (2%) will be administered in the web spaces on either side of the digit, followed by a 2.5-mg intramatrical methotrexate injection into each side of the nail at a point 2.5 mm proximal and lateral to the junction of proximal and lateral nail folds.
  Other Names: Intra-lesional

SUMMARY:
The aim of this study is to compare the efficacy of excimer laser in combination with intralesional MTX injection to intralesional MTX injection alone in treating nail psoriasis

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory disease affecting the skin, nails, and joints. Approximately 61% of psoriatic patients have nail involvement. This percentage can increase up to 90% in patients with psoriatic arthritis. Clinically, nail disease has many presentations depending on the location of the inflammatory process in either the matrix, the nail bed, or the periungual tissue, which results in distinct injury patterns.

Nail psoriasis can lead to impairment in the quality of life and work function due to pain, discomfort, and poor esthetic aspect. Treating nail involvement is important in improving the health outcomes and quality of life among patients with psoriasis. Nail psoriasis is a clinical diagnosis generally made in the context of existing psoriatic skin lesions. The nail psoriasis severity index (NAPSI) has recently been reported as a possible reproducible, objective, and simple tool for clinical assessment of psoriatic nail disease.

Treatment of nail psoriasis is challenging because of the anatomical properties of the nail unit that act as a barrier to active drug delivery and the naturally slow growth rate of the nail plate, which often delays noticeable clinical responses by months. Treatment options available for nail psoriasis include topical therapy, intralesional injections, and systemic and biologic agents. Poor penetration of topical therapy into the nail and surrounding tissue, adverse effects and monitoring of systemic therapies, and patient adherence to therapy make the treatment of nail psoriasis a challenge.

Few publications have been recently concerned intralesional injection of methotrexate in nail psoriasis. This therapy was documented for the first time in 2011. Intramatricial injection of methotrexate is an interesting intralesional therapy as it provides a higher concentration of the drug at the site of action, while avoiding the complications seen with triamcinolone acetonide (injection site atrophy, disappearance of the phalanx under injection, or tendon rupture) The use of excimer laser for the treatment of psoriasis was first documented in 1997. The excimer laser induces T-cell apoptosis characterized by breaks in DNA strands as well as expression of mitochondrial proteins associated with cell death.

ELIGIBILITY:
Inclusion Criteria:

* patients with bilateral fingernail psoriasis will be recruited. The diagnosis will be based upon the clinical characteristics of nail psoriasis.
* Patients will be included after they have stopped any systemic therapy for at least 8 weeks.

Exclusion Criteria:

* Pregnant or lactating woman
* Patients with history of photosensitivity or keloid formation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Modified Nail Psoriasis Severity Index (mNAPSI) | 6 months
  The mNAPSI scores, ranging from 0 to 3 (pitting, onycholysis, and crumbling) depending on the area of the nail involved, will be calculated and digital photographs of the nails will be taken at baseline, monthly till 3 months of treatment, and 6 months after the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Abdel-Moez, MD, Principal Investigator — Assiut University
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No